CLINICAL TRIAL: NCT01800110
Title: Influence of Pomegranate Juice Consumption on the Level of Antioxidants in Breast Milk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0013-13
Record Dates: First submitted 2013-02-19; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Breast Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): label I- 200 cc pomegranate juice once daily for 6 weeks post partum. label II- control group, no placebo is givening.
  Interventions: Dietary Supplement: pomegranate juice

INTERVENTIONS:
Dietary Supplement: pomegranate juice

SUMMARY:
Many medicinal effects of Pomegranate juices are already known. Mainly known for its anti-viral, anti-bacterial and anti-oxide tendency of pomegranate juice.

Many studies which have demonstrated antioxidant activity of pomegranate juice in the blood and blood cells were published.

In addition, published studies have demonstrated the anti-oxidant activity which inhibit the development of atherosclerosis and stroke, even in patients with diabetes, and its effect of decreasing systolic blood pressure in patients with systemic hypertension.

The purpose of the work is to examine the effect of drinking pomegranate juice on the level of anti-oxidants in human breast milk.

DETAILED DESCRIPTION:
the effect of pomegranate juice consumption on breast milk anti oxidants level.

ELIGIBILITY:
Inclusion Criteria:

* lactating woman

Exclusion Criteria:

* pomegranate allergy
* diabetes mellitus
* use of other Dietary Supplement

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
anti oxidant level in human breast milk | at least one year